CLINICAL TRIAL: NCT00394615
Title: Metabolic Imaging: Predicting Histopathologic Response to Preoperative Chemoradiotherapy for Locally Advanced Rectal Cancer
Brief Title: Metabolic Imaging Predict Histopathologic Response to Preop ChemoXRT for Locally Advanced Rectal CA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocol approval expired
Sponsor: Stanford University (Other)
Collaborators: Stanford Cancer Council (Unknown)
Responsible Party: Albert Koong, Stanford University School of Medicine
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REC0001; NCT00394615; REC0001
Record Dates: First submitted 2006-07-05; First posted 2006-11-01 (Estimated); Last update posted 2010-03-29 (Estimated); Status verified 2010-03

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

INTERVENTIONS:
Procedure: Metabolic Imaging

SUMMARY:
In this research study of metabolic imaging in locally advanced rectal cancer, we hope to learn whether new medical imaging technology can help predict the response of rectal cancer to preoperative chemotherapy and radiation therapy. Ultimately we hope this information will in the future help us predict which patients will benefit from more or less aggressive initial therapy for their rectal cancer.

ELIGIBILITY:
Inclusion Criteria:- You must be diagnosed with locally advanced rectal cancer and have chosen treatment with preoperative chemoradiotherapy followed by surgery, which is a standard treatment approach for this disease. Exclusion Criteria:- You are ineligible for this study if you are pregnant or under the age of 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2003-10; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
To learn whether new medical imaging technology can help predict the response of rectal cancer to preoperative chemotherapy and radiation therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Albert Koong, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States